CLINICAL TRIAL: NCT06530095
Title: ''Impact of Early vs. Delayed Prone Positioning on Oxygenation and Mortality in COVID-19 ARDS Patients: A Retrospective Analysis''
Brief Title: We Compared the Covid-19 Acute Respiratory Distress Syndrome (ARDS) Patients Who Applied Prone Positioning for16-24 Hours vs 24-48 Hours
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022/318
Record Dates: First submitted 2024-07-30; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Morality; Oxygenation Indices; Hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Prone Position

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients who have been in prone positioning for 16-24 hours
  Interventions: Other: prone positioning
- Group B: Patients who have been in prone positioning for 24-48 hours
  Interventions: Other: prone positioning

INTERVENTIONS:
Other: prone positioning — prone positioning

SUMMARY:
The goal of this study is to understand if there is any improvement on oxygenation of patients diagnosed with Covid-19 ARDS patients when we extend the duration of prone positioning.

Second outcome of the study is to investigate mortality of patients when we extend the duration of prone positioning.

ELIGIBILITY:
Inclusion Criteria:

COVİD 19 ARDS patients patients who have been intubated for 48 hours and more

Exclusion Criteria:

Pediatric patients Patients who extubated in less than 48 hours Patients with Lung and pleural malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been admitted in ICU and diagnosed with Covid-19 ARDS.
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Oxygen Saturation Index (OSI) | 48 hours
  OSI is calculated by dividing the product of mean airway pressure (MAP) and FiO2 with SpO2
Oxygenation Index | 48 hours
  Oxygenation index is calculated as OI = MAP × Fio2 × 100 / Pao2, where MAP indicates mean airway pressure and Fio2 indicates fraction of inspired oxygen

SECONDARY OUTCOMES:
ICU mortality | 28 days
  mortality rates during patients admission in the ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr Sadi konuk Research and Training hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No